CLINICAL TRIAL: NCT07178665
Title: A Pilot Prospective Trial to Assess the Feasibility of Preoperative Partial Breast Radiation in Breast Cancer Patients
Brief Title: Pilot Trial of Preop Partial Radiation in Breast Cancer Patients
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: 10th patient enrolled; interim analysis to be completed by HROC after 3-month follow-up completed for the 10th patient enrolled.
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Nisha Ohri, MD, Associate Professor of Radiation Oncology, Rutgers Robert Wood Johnson Medical School, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 152502
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Early-stage Breast Cancer; Breast Carcinoma; DCIS
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Preoperative Partial Breast Irradiation (Experimental): Patients will receive 5 fractions of accelerated partial breast irradiation (APBI) delivered before surgery. Surgery is scheduled 1-3 weeks after radiation. If surgical pathology indicates, additional whole-breast or lymph node radiation may be given postoperatively (3-8 weeks after surgery).
  Interventions: Radiation: Radiation: Accelerated Partial Breast Irradiation (APBI)

INTERVENTIONS:
Radiation: Radiation: Accelerated Partial Breast Irradiation (APBI) — Radiation: Accelerated Partial Breast Irradiation (APBI) - 5 fractions delivered every other day before surgery.
  Procedure: Surgery - lumpectomy or mastectomy scheduled 1-3 weeks after RT; additional whole-breast/lymph node RT if indicated.

SUMMARY:
The purpose of our study is to assess the feasibility of preoperative partial breast (APBI) radiation in breast cancer patients. The primary outcome is the acute wound complication rate. We also aim to evaluate cosmetic outcomes and late toxicities as secondary objectives. Another goal is to examine the histopathology of tumors before and after radiation to assess the response and other immunologic and/or molecular changes to the tumor and its environment elicited by the radiation treatment. We hope that this will guide future trials that could change practice in specific patient subgroups.

DETAILED DESCRIPTION:
Our primary objective is to demonstrate that the incidence of grade 3 or more wound complications in patients with non-metastatic and clinically node negative breast cancer or DCIS who are eligible for BCS and treated with pre-operative partial breast irradiation (PBI) at 1 month is no worse than the rates in the current standard of care (6-20%). Our secondary objective is to demonstrate that the physician reported cosmetic outcome at 1 and 3 years after the end of treatment is better than what has been reported for the current standard of practice for patients undergoing BCS and hypofractionated WBI (around 35% reported poor/fair cosmesis at 3 years, Shaitelman et al.). Tertiary objectives are to measure acute and late radiation-related toxicities, such as radiation dermatitis, telangiectasia, and fibrosis, in this cohort of patients and to measure biologic markers that radiation may influence.

To measure the pre-operative APBI clinical target volume (CTV) and compare it to the post-op APBI CTV volume that would have been contoured as CTV if the partial breast was to be delivered post-operatively.

To measure the incidence of fair/poor patient-reported cosmetic outcomes using the BCTOS cosmetic scale.

To study cancer biology before and after radiation treatment.

ELIGIBILITY:
Inclusion Criteria:

Breast cancer patients with biopsy-proven invasive ductal cancer or DCIS Tumor size ≤ 2cm clinically and radiographically Estrogen-receptor positive (ER+) on biopsy Grade 1 or 2 on biopsy Clinically and radiographically node-negative disease No indication of metastatic disease Age >50 Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1 Negative serum pregnancy test if applicable Willingness to participate in the clinical trial and adhere to the study protocol Ability to understand and consent to the study

Exclusion Criteria:

Indication for neoadjuvant chemotherapy or hormone therapy Tumor size >2cm clinically or radiographically ER- on biopsy G3 invasive cancer or DCIS on biopsy Lobular histology Multicentric/multifocal tumor BRCA+ gene mutation Prior ipsilateral breast or thoracic RT Contraindication for baseline MRI Contraindication for surgery Distant metastatic disease Other synchronous cancer (besides bilateral breast) Contraindication to Radiation therapy (presence of scleroderma or other collagen vascular disease) Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Safety and feasibility of preoperative APBI | Up to 30 days after surgery (with continued safety monitoring through 3 years).
  Evaluate the rate of surgical wound complications (infection, delayed healing, dehiscence) following preoperative accelerated partial breast irradiation (APBI).

SECONDARY OUTCOMES:
Quality of life (QoL) | At consultation, and selected follow-up visits up to 3 years.
  Patient-reported outcomes from QoL questionnaires about well-being and treatment experience.

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - RWJBarnabas Health Clara Maas Medical Center, Belleville, New Jersey
  - Trinitas Hospital and Comprehensive Cancer Center, Elizabeth, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital, Hamilton, Hamilton, New Jersey
  - RWJBarnabas Health Jersey City Medical Center, Jersey City, New Jersey
  - Cooperman Barnabas Medical Center, Livingston, New Jersey
  - RWJBarnabas Health - Monmouth Medical Center, Long Branch, New Jersey
  - Jack and Sheryl Morris Cancer Center, New Brunswick, New Jersey
  - RWJBarnabas Health Newark Beth Israel Medical Center, Newark, New Jersey
  - RWJBarnabas Health - Robert Wood Johnson University Hospital Somerset, Somerset, New Jersey
  - RWJBarnabas Health - Community Medical Center, Toms River, New Jersey

IPD SHARING:
Plan to Share IPD: No